CLINICAL TRIAL: NCT01379729
Title: Functional Survival of Beta Cell Allografts After Transplantation in the Peritoneal Cavity of Non-uremic Type 1 Diabetic Patients
Brief Title: Bet Cell Therapy in Diabetes Type 1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ-VUB (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Bart Keymeulen, MD. PhD., AZ-VUB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK_TX_07
Record Dates: First submitted 2011-05-02; First posted 2011-06-23 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Transplantation; Beta Cells; Encapsulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Patients with loss of long-term function after intraportal implantation
  Interventions: Other: Transplantation of encapsulated beta cells.
- Group B (Active Comparator): Patients that are candidates for islet cell transplantation
  Interventions: Other: Transplantation of encapsulated beta cells.

INTERVENTIONS:
Other: Transplantation of encapsulated beta cells. — Implantation of a therapeutical dose of encapsulated beta cells.
  Other Names: encapsulated beta cells
  Arms: Group A
Other: Transplantation of encapsulated beta cells. — Implantation of a therapeutical dose of encapsulated beta cells.
  Other Names: encapsulated beta cells
  Arms: Group B

SUMMARY:
Primary outcome measurement is a parameter of functional beta cell mass at 6 months PT. Functional beta-cell mass will be calculated using the AUC/min between 150 and 160 min during hyperglycemic clamp at 180 mg/dl.

The investigators hypothesize that functional beta-cell mass will be more than 20% compared to healthy controls.

Secondary outcome measurements:

Functional beta-cell mass at 2,12,18,24,36,48 and 60 months PT.

The investigators will also compare at 2, 6,12, 24,36,48 and 60 months the changes against base-line (base-line = before first intraperitoneal transplantation):

* metabolic control
* safety parameters
* episodes of hypoglycemia
* islet cell autoantibodies, lymphocyte subsets, T-cell reactivity against auto- and alloantigens using pre-transplant measurements as base-line The investigators hypothesize that metabolic control and prevalence of hypoglycemia, will be significantly improved till PT month 12.

Histopathology of a biopsy specimen of the human intraperitoneal beta cell implant, at time of the second implant. Comparison with composition of graft, identification of microenvironment of host origin and correlation with functional assessment will be performed.

DETAILED DESCRIPTION:
In recipients with loss of long-term function after intraportal implantation (Group A)

1. To implant an alginate embedded human beta cell graft in a "therapeutic" dose in the intraperitoneal cavity of type 1 diabetic patients under immunosuppression with tacrolimus/MMF.
2. To obtain histopathology of a biopsy specimen of the intraperitoneal human beta cell implant.
3. To assess the safety profile, metabolic and immune effects of alginate embedded implants in the intraperitoneal cavity.

   In patients that are candidates for islet cell transplantation (Group B)
4. To implant an alginate embedded human beta cell graft in a "therapeutic" dose in intraperitoneal cavity of type 1 diabetic patients under immunosuppression with tacrolimus/MMF.
5. To obtain histopathology of a biopsy specimen of the intraperitoneal human beta cell implant
6. To assess the safety profile, metabolic and immune effects of alginate embedded implants in the intraperitoneal cavity.

ELIGIBILITY:
Inclusion Criteria:

Group A:

Patients with loss of long-term function after intraportal implantation (- Patients with type 1 insulin-dependent diabetes who received two intraportal implantations > 12 months ago.

* Random C-peptide between 0.09 and 0.5 ng/dl (glycemia between 100 and 200 mg/dl)
* Cooperative and reliable patient giving informed consent by signature

Group B:

Patients that are candidates for islet cell transplantation - age 18-65 years, male or female, Caucasian or not; only subjects < 50 yrs will be allocated to the rituximab treatment arm

* body weight < 100 kg; patients with a bodyweight of < 80kg, will receive priority
* patients with a BMI ≤ 27 kg/m2 will receive priority
* Type 1 insulin-dependent diabetes
* C-peptide < 0.07 nmol/l (< 0.2 µg/l) 6 min. after glucagon IV (1mg) (glycemia > 180 mg/dl)
* Intensive insulin therapy for more than two years, patients with insulin pump during at least 2 months before inclusion will receive priority
* Patients should have at least one of the following chronic complications of diabetes:

  * albuminuria 30-1000mg/ 24hrs on 3 separate determinations (>1 month) outside an episode of illness, despite intake of ACE inhibitors; mean systolic blood pressure should be under 130 mmHg and mean diastolic blood pressure under 85 mmHg, when measured at home with ambulatory BP monitoring
  * moderate or severe non-proliferative or proliferative retinopathy
  * hypoglycemic unawareness
* Cooperative and reliable patient giving informed consent by signature

Exclusion Criteria:

* Women of reproductive age

  * Smoker
  * EBV antibody negativity
  * HIV 1 & 2 antibody positivity
  * CMV IgM positivity
  * Hepatitis B infection
  * GFR < 45 ml/min/1.72 m2
  * Albuminuria ≥ 1000 mg/24 hrs
  * History of thrombosis or pulmonary embolism
  * History of malignancy, tuberculosis or chronic viral hepatitis
  * History of any other serious illness which could be relevant for the protocol
  * Presence of clinical significant HLA antibodies
  * Blood donation within one month prior to screening
  * Symptoms and/or signs of infection, particularly (present or past) endocarditis, osteomyelitis
  * Any history of hepatic or neoplastic disease
  * Any history of renal disease (except diabetes)
  * Abnormal liver function tests and/or NMR of liver
  * Hemoglobinopathy
  * History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the patient
  * Use of illicit drugs or overconsumption of alcohol (> 3 IU/day) or history of drug or alcohol abuse
  * Being legally incapacitated, having significant emotional problems at the time of the study, or having a history of a psychiatric disorder that may be exacerbated by the transplantation procedure or interfere with compliance during follow-up
  * Having received antidepressant medications during the last 6 months
  * Participating in another pharmacological study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measurement is a parameter of functional beta cell mass at 6 months PT. Functional beta-cell mass will be calculated using the AUC/min between 150 and 160 min during hyperglycemic clamp at 180 mg/dl. | 6 months PT.

SECONDARY OUTCOMES:
Functional beta-cell mass at 2,12,18,24,36,48 and 60 months PT. | 60 months
  Functional beta-cell mass at 2,12,18,24,36,48 and 60 months PT.
  The investigators will also compare at 2, 6,12, 24,36,48 and 60 months the changes against base-line (base-line = before first intraperitoneal transplantation):
  * metabolic control
  * safety parameters
  * episodes of hypoglycemia
  * islet cell autoantibodies, lymphocyte subsets, T-cell reactivity against auto- and alloantigens using pre-transplant measurements as base-line
Functional beta-cell mass at 2,12,18,24,36,48 and 60 months PT. | 60 months
  Functional beta-cell mass at 2,12,18,24,36,48 and 60 months PT.
Changes from Baseline | 60 months
  The investigators will also compare at 2, 6,12, 24,36,48 and 60 months the changes against base-line (base-line = before first intraperitoneal transplantation):
  * metabolic control
  * safety parameters
  * episodes of hypoglycemia
  * islet cell autoantibodies, lymphocyte subsets, T-cell reactivity against auto- and alloantigens using pre-transplant measurements as base-line

CONTACTS AND LOCATIONS:
Overall Officials: Bart Keymeulen, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - UZ Brussel, Brussels
  - UZ Leuven, Leuven

REFERENCES:
- [Background] Gillard P, Keymeulen B, Mathieu C. Beta-cell transplantation in type 1 diabetic patients: a work in progress to cure. Verh K Acad Geneeskd Belg. 2010;72(1-2):71-98. PMID 20726441
- [Background] Hilbrands R, Huurman VA, Gillard P, Velthuis JH, De Waele M, Mathieu C, Kaufman L, Pipeleers-Marichal M, Ling Z, Movahedi B, Jacobs-Tulleneers-Thevissen D, Monbaliu D, Ysebaert D, Gorus FK, Roep BO, Pipeleers DG, Keymeulen B. Differences in baseline lymphocyte counts and autoreactivity are associated with differences in outcome of islet cell transplantation in type 1 diabetic patients. Diabetes. 2009 Oct;58(10):2267-76. doi: 10.2337/db09-0160. Epub 2009 Jul 14. PMID 19602536
- [Background] Gillard P, Vandemeulebroucke E, Keymeulen B, Pirenne J, Maes B, De Pauw P, Vanrenterghem Y, Pipeleers D, Mathieu C. Functional beta-cell mass and insulin sensitivity is decreased in insulin-independent pancreas-kidney recipients. Transplantation. 2009 Feb 15;87(3):402-7. doi: 10.1097/TP.0b013e3181928a1c. PMID 19202446
- [Background] Pipeleers D, Chintinne M, Denys B, Martens G, Keymeulen B, Gorus F. Restoring a functional beta-cell mass in diabetes. Diabetes Obes Metab. 2008 Nov;10 Suppl 4:54-62. doi: 10.1111/j.1463-1326.2008.00941.x. PMID 18834433
- [Background] Keymeulen B. Therapies aimed at preservation or restoration of beta cell function in type 1 diabetes. Verh K Acad Geneeskd Belg. 2008;70(2):85-103. PMID 18630722
- [Derived] Jacobs-Tulleneers-Thevissen D, Chintinne M, Ling Z, Gillard P, Schoonjans L, Delvaux G, Strand BL, Gorus F, Keymeulen B, Pipeleers D; Beta Cell Therapy Consortium EU-FP7. Sustained function of alginate-encapsulated human islet cell implants in the peritoneal cavity of mice leading to a pilot study in a type 1 diabetic patient. Diabetologia. 2013 Jul;56(7):1605-14. doi: 10.1007/s00125-013-2906-0. Epub 2013 Apr 26. PMID 23620058